CLINICAL TRIAL: NCT04872530
Title: Bioavailability of Amino Acids and Metabolic Products Following Oral Ingestion of Plant-Based Proteins in Young, Healthy Men and Women Aged 18-35y
Brief Title: Bioavailability of Plant Protein Amino Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Marigot Ltd. (Industry); Enterprise Ireland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019_12_02_EHS
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Bioavailability of Amino Acids Following Oral Ingestion of Plant-Based Proteins in Young, Healthy Men
Keywords: Bioavailability of Amino Acids Following Oral Ingestion of Plant-Based Proteins in Young, Healthy Men
MeSH Terms: interventions — Whey

STUDY DESIGN:
Intervention Model Description: Subjects who volunteer for this study will undertake SIX controlled feeding trials, each trial separated by 7 days.Subjects will be assigned to a randomised sequence of six protein isolates including: (1) pea-protein concentrate; (2) fava-bean protein concentrate; (3) chickpea protein concentrate; (4) red lentil protein concentrate; (5) non-essential amino acid blend (negative control);( 6) whey protein concentrate. Protein is dosed at 0.33 g/kg body mass in 500 ml of water.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pea-protein concentrate (Experimental): Pea-protein concentrate dosed at 0.33 g/kg body mass in 500 ml of water.
  Interventions: Dietary Supplement: Pea-protein concentrate
- Fava-bean protein concentrate (Experimental): Fava-bean protein concentrate dosed at 0.33 g/kg body mass in 500 ml of water.
  Interventions: Dietary Supplement: Fava-bean protein concentrate
- Chickpea protein concentrate (Experimental): Chickpea protein concentrate dosed at 0.33 g/kg body mass in 500 ml of water.
  Interventions: Dietary Supplement: Chickpea protein concentrate
- Red lentil protein concentrate (Experimental): Red lentil protein concentrate dosed at 0.33 g/kg body mass in 500 ml of water.
  Interventions: Dietary Supplement: Red lentil protein concentrate
- Non-essential amino acid blend (Experimental): Non-essential amino acid blend dosed at 0.33 g/kg body mass in 500 ml of water.
  Interventions: Dietary Supplement: Non-essential amino acid blend
- Whey protein concentrate (Experimental): Whey protein concentrate dosed at 0.33 g/kg body mass in 500 ml of water.
  Interventions: Dietary Supplement: Whey protein concentrate

INTERVENTIONS:
Dietary Supplement: Pea-protein concentrate — Pea-protein concentrate
  Arms: Pea-protein concentrate
Dietary Supplement: Fava-bean protein concentrate — Fava-bean protein concentrate
  Arms: Fava-bean protein concentrate
Dietary Supplement: Chickpea protein concentrate — Chickpea protein concentrate
  Arms: Chickpea protein concentrate
Dietary Supplement: Red lentil protein concentrate — Red lentil protein concentrate
  Arms: Red lentil protein concentrate
Dietary Supplement: Non-essential amino acid blend — Non-essential amino acid blend
  Arms: Non-essential amino acid blend
Dietary Supplement: Whey protein concentrate — Whey protein concentrate
  Arms: Whey protein concentrate

SUMMARY:
This study aims to inform of the mechanism of action of plant-based protein by measuring the bioavailability (i.e. rate of appearance and magnitude of concentration in the circulation following oral ingestion) of key amino acid and metabolic products that regulate skeletal muscle protein synthesis (MPS) in humans.

DETAILED DESCRIPTION:
Plant-based proteins contain several amino acids that are essential to signal muscle growth/repair and act as a substrate during muscle protein synthesis. However, compared to animal protein or free-amino acids, the bioavailability of certain essential amino acids may be compromised. Following selective processing (e.g. removal of carbohydrate and/or other anti-nutritive factors) food grade plant-based protein concentrates possibly confer greater bioavailability and bioactivity in vivo. This project explores the bioavailability and bioactivity of selected plant-based protein concentrates following oral ingestion in young, healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* No known intolerance to any item contained in the protein products.
* No blood borne disease risk, current illness or medication that would adversely affect participation
* No known adverse reaction to venepuncture

Exclusion Criteria:

* n/a

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy young men
Enrollment: 10 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Plasma amino acids | 3 hours
  Plasma amino acids measured by HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Phil Jakeman, PhD, Principal Investigator — University of Limerick
Locations (1):
- Education and Health Sciences, Limerick, Ireland